CLINICAL TRIAL: NCT00662285
Title: Description of Iron Status in Blood Donors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Haukeland University Hospital (Other)
Responsible Party: Haukeland University Hospital and University of Bergen, Blood bank and Institute of medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 16225
Record Dates: First submitted 2008-04-16; First posted 2008-04-21 (Estimated); Last update posted 2008-04-21 (Estimated); Status verified 2008-04

CONDITIONS: Iron Deficiency
Keywords: iron status; blood donors
MeSH Terms: conditions — Iron Deficiencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A: Niferex (Other): 100 mg Fe++
  Interventions: Dietary Supplement: Iron supplement: Niferex 100 mg

INTERVENTIONS:
Dietary Supplement: Iron supplement: Niferex 100 mg — A: 100 mg pr day in 8 days

SUMMARY:
Description of the effect of standard iron supplement on iron status in blood donors

Hypothesis:

For each person in each group (group a "without iron supplement" or group b "with iron supplement") individual biological variation in reticulocytes, tested day 1 and day 8 will be described. Groups a and b will be compared on iron status from day 1 and day 8.

* H1 null: There is no significant intraindividual difference in reticstatus at day 1 and at day 8, in group a.
* H2 null: There is no significant intraindividual difference in reticstatus at day 1 and at day 8, in group b
* H3 null: There is no significant difference in iron status for the two groups, a and b, at day 1 and at day 8.

DETAILED DESCRIPTION:
The purpose of the study:

The purpose of the study is to describe intra- individual biological variation in reticulocyte parameters in established blood donors. The aim is also to compare iron status and reticulocyte parameters in a group of established donors who are offered iron supplement, to a comparable group who are not offered iron supplement, at the time of donation and one week after donation.

Design:

The design is a prospective longitudinal intervention-study, with randomised subjects to iron supplement/ not iron supplement groups.

Materials and methods:

Each subject will be tested with an extended test repertoire at the time of donation, day one, and the same test repertoire will be repeated one week after donation, day eight. Iron supplement is defined as100 mg of iron-sulphate (Ferro retard), taken once a day. Subjects are randomised into two groups; group a: "no iron supplement", n = 100, and group b: "iron supplement", n = 100. These groups will be stratified according to gender and age. Randomising will be done without knowledge of earlier blood tests. Subjects are asked to participate as they arrive for blood donation, by oral and written information. Questionnaire for established donors are used at day one. Day eight, follow-up of iron supplements will be controlled.

Dropouts and withdrawal:

Subjects who do not receive iron supplement are at risk of developing iron deficiency. Criteria for transfer to treatment group will be:

* Females: Hb < 12.5 g/dL
* Males: Hb < 13.5 g/dL These subjects may continue as participants in the study, but with a description of transfer to treatment group including date and treatment type (iron supplement type and dose, dose interval, treatment time, termination of treatment).

Ethics:

The study is approved by the regional ethics committee. All subjects must sign informed consent.

Data analysis:

Univariate and multivariate analysis are use for iron status variables, with separate analysis for each gender. Baseline data are taken at day one, at donation, and follow up testing at day eight. Dependent variables are haemoglobin, S-ferritin, total reticulocytes count, haemoglobin content in reticulocytes and percent hypochromated red cells. Independent variables are gender, age, ironsupplement/ no iron supplement.

Biochemical tests:

Test methods are specified, and instruments described. Biochemical test are performed at lab for clinical biochemistry, Haukeland University Hospital, Bergen.

ELIGIBILITY:
Inclusion Criteria:

* Must be accepted as blood donor

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2008-04; Primary Completion 2008-04 (Estimated); Study Completion 2009-04 (Estimated)

PRIMARY OUTCOMES:
Iron status | april 2008

SECONDARY OUTCOMES:
Hemoglobin and serum ferritin | april 2008

CONTACTS AND LOCATIONS:
Overall Officials: Anne S Røsvik, Study Chair — Aalesund University College
Locations (2):
- Norway (2):
  - Blood bank, Haukeland University Hospital,, Bergen
  - Blood bank, Bergen